CLINICAL TRIAL: NCT00175383
Title: A Randomized Trial of Short Versus Long Acting LHRH Agonist Preparation Prior to Transperineal Implantation of the Prostate
Brief Title: Long Acting LHRH Versus Short Acting LHRH in the Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03-1213
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer, LHRH, hormone therapy, testosterone level
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leuprolide preparations (Experimental): One versus three-month Leuprolide preparations in patients otherwise suitable for our Brachytherapy Program
  Interventions: Drug: luteinizing hormone-releasing hormone (LHRH) short acting or long acting

INTERVENTIONS:
Drug: luteinizing hormone-releasing hormone (LHRH) short acting or long acting — See Detailed Description.

SUMMARY:
Brachytherapy, or Transperineal implantation of the prostate (TPIP), is a recognized form of treatment for localized cancer of the prostate. TPIP has been used at the British Columbia Cancer Agency (BCCA) since 1998. As part of the treatment, some patients also require hormone therapy for 6 months. This is given as injections of a drug called an LHRH agonist. The LHRH agonist is made either as short-acting (1-month) or long-acting (3 month) injections. The LHRH agonist lowers testosterone levels, which helps make delivery of TPIP easier, and more effective.

There are specific guidelines regarding the use of LHRH agonist treatment with brachytherapy, however there is no policy whether short-acting or long-acting LHRH agonists should be used.

Analysis of results from BC has shown that there seems to be a delay in the time in which testosterone levels return to normal in men who receive the long-acting LHRH agonist compared with the short-acting LHRH agonist, however this is not known for sure.

DETAILED DESCRIPTION:
The suppression of testosterone to castrate levels has a definite advantage in terms of prostate volume downsizing, disease control and ease of Brachytherapy, in this patient population. The improved potency preservation rate seen with brachytherapy, when compared to other treatments such as radical prostatectomy or external beam, may be an important determinant in the patient's choice of treatment modality. Hence, testosterone recovery should be an important endpoint to consider in this patient population since prolongation of testosterone suppression may also delay the return of erectile function.

In order to compare the impact of LHRH agonist preparations on the rate of testosterone recovery, we propose a randomized clinical trial using one versus three-month Leuprolide preparations in patients otherwise suitable for our Brachytherapy Program.

The primary objective of this study is the median time to testosterone recovery in patients receiving 6 X 1-month or 2 X 3-month LHrH preparations and TPIP as radical treatment for limited stage prostate cancer.

In this context, testosterone recovery is defined as the return to the lower limit of normal for the patient's age group as well as return to pre treatment levels.

Analysis will mainly focus on time to testosterone recovery as defined by return to the lower limit of normal for the patient's age group as well as return to pre treatment levels. The lower limits of normal are defined as 5.8nmol/L and 5.5nmol/L for < 50 and > 50 years old

Changes in PSA level, QOL and erectile function will also be recorded

ELIGIBILITY:
Inclusion Criteria:

All patients who elect to undergo brachytherapy for the treatment of adenocarcinoma of the prostate and who are otherwise recommended treatment with LHRH agonist. All patients must have a confirmed histological diagnosis of adenocarcinoma of the prostate and elect to be treated with transperineal implantation of the prostate.

Eligible patients will have confirmed clinical stage T1 or T2 (UICC 1997 staging system) with

1. PSA > 10 but < 15 and Gleason score < 7, OR
2. PSA < 10 and Gleason score = 7 OR
3. Prostate volume > 50cc as measured on trans rectal ultrasound

While criteria 1 and 2 are mutually exclusive, criteria 3 can be present alone or in combination with criteria 1 OR 2.

Otherwise patients should be able to give informed consent and have a life expectancy. 2 years.

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is the median time to testosterone recovery in patients receiving 6 X 1-month or 2 X 3-month LHrH preparations and TPIP as radical treatment for limited stage prostate cancer. | 6 months
In this context, testosterone recovery is defined as the return to the lower limit of normal for the patient's age group as well as return to pre treatment levels.

SECONDARY OUTCOMES:
PSA profile, quality of life, sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Eric Berthelet, MD, Principal Investigator — The University of British Columbia
Locations (1):
- BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia, Canada